CLINICAL TRIAL: NCT06463340
Title: A First-In-Human, Phase 1, Dose Escalation Study of SGR-3515 In Participants With Advanced Solid Tumors.
Brief Title: Study of SGR-3515 In Participants With Advanced Solid Tumors.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Schrödinger, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGR-3515-101
Record Dates: First submitted 2024-05-24; First posted 2024-06-17 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumor
Keywords: Solid Tumor; Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation (Experimental): 28-day treatment cycle.
  Interventions: Drug: SGR-3515

INTERVENTIONS:
Drug: SGR-3515 — SGR-3515 will be administered orally with an intermittent schedule.

SUMMARY:
The purpose of this study is to learn about the effects of a new study drug, called SGR-3515 that may be a treatment for advanced solid tumors.

DETAILED DESCRIPTION:
SGR-3515-101 is a phase 1, first-in-human, single agent, dose-escalation study designed to evaluate the safety, tolerability, dose limiting toxicities, pharmacokinetics, pharmacodynamics, and preliminary anti-tumor activity of SGR-3515 and to identify the maximum tolerated dose, recommended phase 2 dose and schedule of SGR-3515, in participants with advanced solid tumors hypothesized to be sensitive to Wee1/Myt1 inhibition and any solid tumors with designated molecular perturbation relevant to DNA damage repair pathway, including but not limited to CCNE1 amplification.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced/metastatic solid tumor
* Measurable disease per RECIST version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Participant must understand and sign an Informed Consent Form (ICF) prior to any study-related assessments/procedures
* Adequate bone marrow and organ function
* Women of child-bearing potential (WOCBP) or males must agree to use highly effective contraception for the duration of study and for 90 days after the last dose of study drug

Exclusion Criteria

* Participants with primary Central Nervous System (CNS tumors).
* Participant has received prior systemic anti-cancer treatments or other investigational agents ≤ 21 days of first dose of study drug, or 5 half-lives, whichever is shorter
* Participant who has received definitive local control radiation (any dose greater than 50 Gy) < 42 days prior to the first dose of study drug.
* Participant who has received major surgeries ≤ 21 days prior to first dose of study drug
* Participants who have not recovered to Grade 1 or baseline levels from toxicity or adverse events related to prior treatment for their cancer, excluding Grade 2 alopecia, peripheral neuropathy and ototoxicity.
* Participant who has another clinically significant invasive malignancy, as determined by the investigator, ≤ 2 years prior to the first dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Day 1 to 28 days after the last dose of SGR-3515.
  Incidence and severity of adverse events (AEs) per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0 and changes in hematology and chemistry values, vital signs, electrocardiograms (ECGs); and dose interruptions, dose reductions, dose delays and study drug discontinuation due to AEs.
Incidence of Dose Limiting Toxicities (DLTs) | Day 1 to Day 28 of the first 28-day dosing cycle.
  Incidence of Dose Limiting Toxicities (DLTs)
Incidence of serious adverse events (SAEs) | Day 1 to 28 days after the last dose of SGR-3515
  Incidence of serious adverse events (SAEs)
Recommended phase 2 dose and schedule | From day 1 until end of phase I when Maximum Tolerated Dose (MTD) and schedule has been reached and confirmed.
  Recommended phase 2 dose and schedule

SECONDARY OUTCOMES:
Pharmacokinetics: Measures Cmax and Cmin of SGR-3515 | Day 1 to Day 28 of first 28-day dosing cycle
  Pharmacokinetics: Cmax and Cmin of SGR-3515
Pharmacokinetics Measures: t1/2 of SGR-3515 | Day 1 to Day 28 of first 28-day dosing cycle
  Pharmacokinetics: t1/2 of SGR-3515
Pharmacokinetics Measures: tmax of SGR-3515 | Day 1 to Day 28 of first 28-day dosing cycle
  Pharmacokinetics: tmax of SGR-3515
Pharmacokinetics Measures: Area Under the Curve (AUC) of SGR-3515 | Day 1 to Day 28 of first 28-day dosing cycle
  Pharmacokinetics: Area Under the Curve (AUC) of SGR-3515
Efficacy analysis | Day 1 to end of Phase I study
  Efficacy analysis will be performed for each dose level and include but not limited to objective response rate (ORR), duration of response (DOR), disease control rate (DCR) and duration of disease control (DDC), which will be assessed by investigators

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Dugan, MD, Study Director — CMO/Study Physician
Locations (14):
- United States (13):
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center/Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - NEXT Virginia, Fairfax, Virginia
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada